CLINICAL TRIAL: NCT01571882
Title: Effects of the Consumption of a no Added Sugar Fermented Milk Product Enriched With Plant Sterols and Policosanols on Hypercholesterolaemia Management in Moderately Hypercholesterolaemic Adults
Brief Title: Effects of Fermented Milk Product Enriched With Plant Sterols and Policosanols in Mild Hypercholesterolaemic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: NU235
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Mildly Hypercholesterolemic Subjects
Keywords: Plant sterol - Policosanols - Hypercholesterolemia - Dairy
MeSH Terms: interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 = Tested product 1 (Experimental)
  Interventions: Other: 1- Low fat drinkable fermented dairy product enriched with 1.6g of plant sterol (as free equivalent) + 10 mg of policosanols per unit
- 2 = tested product 2 (Experimental)
  Interventions: Other: 2- Low fat drinkable fermented dairy product enriched with 1.6g of plant sterol (as free equivalent) + 20 mg of policosanols per unit
- 3 = Active control product (Active Comparator)
  Interventions: Other: 3- Low fat drinkable fermented dairy product with 1.6g of plant sterol (as free equivalent) but without policosanols (Active control)

INTERVENTIONS:
Other: 1- Low fat drinkable fermented dairy product enriched with 1.6g of plant sterol (as free equivalent) + 10 mg of policosanols per unit — 1- Intervention with test product ( 1.6g of plant sterol + 10 mg of policosanols/ day)
  Arms: 1 = Tested product 1
Other: 2- Low fat drinkable fermented dairy product enriched with 1.6g of plant sterol (as free equivalent) + 20 mg of policosanols per unit — 2- Intervention with test product (1.6g of plant sterol + 20 mg of policosanols/day)
  Arms: 2 = tested product 2
Other: 3- Low fat drinkable fermented dairy product with 1.6g of plant sterol (as free equivalent) but without policosanols (Active control) — 3- Intervention with active control product (1,6 g of plant sterol/ day)
  Arms: 3 = Active control product

SUMMARY:
The objective of this study is to investigate the effect of consumption of a low-fat, no added sugar, dairy fermented product enriched with plant sterols and policosanols at two doses, on LDL-cholesterol concentration in hypercholesterolaemic adults after 3 weeks of product consumption versus active control product.

ELIGIBILITY:
Inclusion Criteria:

* male and female aged 20-75 years;
* BMI between 19 and 30 kg/m2 ,
* LDL-cholesterol plasma level between 130 mg/dL and 190 mg/dL (bounds included) stabilized for more than 3 months,
* without statin monotherapy or other hypocholesterolaemic drug treatment,
* accepting to follow the dietary recommendations advisable for hypercholesterolemic patient (NCEP-ATP III guidelines)

Exclusion Criteria:

* serum triglyceride (TG) levels ≥ 4 mmol/L (3.5 g/L), having experienced any cardiovascular event in the last 6 months,
* receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-06; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Guildford Clinical Pharmacology Unit Ltd. (Gcpl), Guildford, Surrey, United Kingdom